CLINICAL TRIAL: NCT04573959
Title: Validation of CapsoVision CapsoCam® SV-3 Capsule Endoscopy System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capso Vision, Inc. (Industry)
Collaborators: Generic Devices Consulting, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CVI-006
Record Dates: First submitted 2020-02-07; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Intestinal Disease; Inflammatory Bowel Diseases; Crohn Disease; Ulcer; Celiac Disease
Keywords: Intestinal Disease; Inflammatory Bowel Diseases; Crohn Disease; Ulcer; Celiac Disease; Angioectasia; Polyp
MeSH Terms: conditions — Intestinal Diseases; Inflammatory Bowel Diseases; Crohn Disease; Ulcer; Celiac Disease; Polyps | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- SV-3 Capsule Endoscopy (Experimental): CapsoCam SV-3 Capsule Endoscopy system will perform in a manner consistent with the performance of the CapsoCam SV-3 capsule endoscopy systems.
  Interventions: Device: SV-3 Capsule Endoscopy

INTERVENTIONS:
Device: SV-3 Capsule Endoscopy — The purpose of this study is to validate an updated version of the CapsoCam SV-3 Endoscopy System with respect to the reproducibility of the system to capture and download small bowel images in a manner consistent with the predicate CapsoCam SV-3 capsule endoscopy.
  Other Names: Capsule Endoscopy System

SUMMARY:
To validate an updated version of CapsoCam® SV-3 Endoscopy System brand name CapsoCam Plus™) with respect to the reproducibility of the system to capture and download small bowel images in a manner consistent with the predicate CapsoCam® SV-2 and SV-3 capsule endoscopy systems.

DETAILED DESCRIPTION:
The purpose of the study is validate the an updated version of the CapsoCam® SV-3 Endoscopy System brand name CapsoCam Plus™) with respect to the reproducibility of the system to capture and download small bowel images in a manner consistent with the predicate CapsoCam® SV-2 and SV-3 capsule endoscopy systems.

The system to be validated consists of an updated version of the CapsoCam® SV-3 video capsule endoscope, the CapsoView® CVV Software, the CapsoAccess ® Capsule Data Access System (CDAS3) and the CapsoRetrieve® Capsule Retrieval Kit for the collection of the excreted CapsoCam capsule.

The captured CapsoCam® SV-3 capsule images of the small bowel will be downloaded via the CapsoAccess® Capsule Data Access System (CDAS3) to a computer and proprietary CapsoView® CVV Software is used to review capsule images. The CapsoView® software displays the video and employs a variety of image-enhancement, video playback, and image analysis features to facilitate physician review of the captured images. The software allows the physician to efficiently annotate individual frames from the video and compile a procedure report, which aids in diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Willing and able to provide written informed consent
* Completion of pre-study questionnaire
* Approval of study principal investigator

Exclusion Criteria:

* Subjects with abdominal pain of unknown origin
* Difficulty Swallowing
* Known or suspected gastrointestinal disease
* Diarrhea or constipation
* Anemia of unknown origin
* Rectal or other gastrointestinal bleeding
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

PRIMARY OUTCOMES:
Ability to capture images | 2 weeks
  Images are captured throughout an entire small bowel exam, with complete small bowel exam defined as the ability of the capsule to reach the cecum while still recording images.
Ability to download images | 2 weeks
  Images are correctly downloaded using the CapsoAccess Capsule Data Access System (CDAAS3).
Diagnostic Quality of Images | 2 weeks
  Small bowel images of diagnostic quality are able to be reviewed using the CapsoView CVV Software and determined to be effective for diagnostic purposes by the study investigator.

CONTACTS AND LOCATIONS:
Overall Officials: David Shields, MD, Principal Investigator — CapsoVision Research Center
Locations (1):
- CapsoVision, Inc., Saratoga, California, United States

IPD SHARING:
Plan to Share IPD: No